CLINICAL TRIAL: NCT04221659
Title: Effects of Neuromodulation on Brain Electric Activity of Parkinson's Disease Patients: Randomized Controlled Trial
Brief Title: Effects of Neuromodulation on Brain Electric Activity of Parkinson's Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator and Teacher, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EEGPark
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS over M1 and DLPFC (Experimental): Anodic transcranial direct current stimulation (tDCS) over right primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation
- tDCS over M1 and FPA (Experimental): Anodic transcranial direct current stimulation (tDCS) over right primary motor cortex (M1) and left frontal polar area (FPA). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation
- tDCS over M1 (Active Comparator): Anodic transcranial direct current stimulation (tDCS) over right primary motor cortex (M1). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Participants will receive 16 sessions of Transcranial Direct Current Stimulation (tDCS) for 20 minutes each at 2 mA intensity, on alternate days (3 times a week). The current will be delivered via saline-embedded sponge surface electrodes using a battery-powered neurostimulator (TCT-Research, Trans Cranial Technologies, Hong Kong). A small active specific electrode (5x5 cm) will be used to prevent coverage of adjacent areas, resulting in a current density of 0.08 mA / cm². The cathode, reference electrode (5x7cm), will be positioned in the occipital region. These parameters are within the safe limits established in previous human studies.

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative and progressive movement disorder, whose population incidence is increasing. It is characterized by motor symptoms such as tremor, stiffness and bradykinesia, and non-motor symptoms, highlighting the executive dysfunction that can be present from the early stages of the disease. These deficits increase the risk of falls and reduce functional independence. Transcranial Direct Current Stimulation (ETCC) can be an attractive rehabilitation option in PD because it is a non-invasive and safe method that can modulate cortical excitability and improve motor and non-motor symptoms. One of the techniques to detect neurophysiological biomarkers associated with changes in the functional health of the brain and the effectiveness of this type of treatment is the analysis of microstates from the electroencephalogram (EEG). So, the objective of the present study is to investigate the effects of different assemblies of multifocal ETCC on the electrical brain activity represented by the EEG microstates and clinical characteristics in patients with PD.

DETAILED DESCRIPTION:
For this, a randomized, triple-blind clinical trial will be conducted with 60 people with PD, between 40 and 75 years old, regardless of sex, recruited from the reference centers in neurology and physiotherapy in João Pessoa-PB. Participants will be randomized into three groups: Group 1 - ETCC over M1 + CPFDL; Group 2 - ETCC on M1 + APF; Group 3 - ETCC on M1. In each condition an initial baseline assessment (T0) will be performed after 16 treatment sessions (T1) and 30 days after the end of the protocol (Follow-up Assessment - T2). The evaluated outcomes will be: analysis of microstates and spectral analysis of frequencies by EEG; dual task capability with Timed Up and Go (TUG); executive function (Stroop test and verbal fluency test); motor aspects of daily life (MDS UPDRS II). For all analyzes, the statistical software SPSS (SPSS Inc, Chicago IL, USA) for Windows, Version 20.0, will be used and statistical significance considered at 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD, issued by a neurologist specializing in movement disorders;
* Disease staging between I and III, according to the modified Hoehn and Yahr scale;
* Regular antiparkinsonian pharmacological treatment;
* Score higher than 24 or 18 (for participants with low education) in the Mini -Mental State Examination

Healthy Subjects inclusion criteria:

* Ages: 40 - 75 years
* Sex: All
* Subjects who do not have self-report of neurodegenerative disorders

Exclusion Criteria:

* Diagnosis of atypical parkinsonism;
* Neurological comorbidities;
* History of epilepsy, neurosurgery (including metal clip implantation) and pacemaker implantation;
* DBS implantation - deep brain stimulation;
* Patients missing two consecutive protocol sessions.

Healthy Subjects exclusion criteria:

* History of epilepsy;
* Metallic implants in the head;
* Clinical evidence of brain injury.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in EEG microstates | Baseline, after 6 weeks, and after 10 weeks
  For the analysis of the EEG microstates the following temporal parameters will be considered: the average duration of each microstate; its frequency of occurrence; the fraction of the total recording time covered by each; the overall variation explained by each microstate and the probabilities of transition from one microstate to another.
  The brain electrical activity will be acquired through the BrainVision actiCHamp equipment using 32 Ag / AgCl electrodes that will be fixed according to the International 10-20 System, keeping the impedance below 10kΩ in silent condition and in eyes open states. and eyes closed. The output of the amplifier data will be directed to a computer with BrainVision Pycoder software to record the obtained records and the data will be processed using the BrainVision Analyzer.

SECONDARY OUTCOMES:
Spectral analysis of EEG frequencies | Baseline, after 6 weeks, and after 10 weeks
  Analyze the average of the spectra in the different frequency bands and identify their predominant cortical regions.
  The brain electrical activity will be acquired through the BrainVision actiCHamp equipment using 32 Ag / AgCl electrodes that will be fixed according to the International 10-20 System, keeping the impedance below 10kΩ in silent condition and in eyes open states. and eyes closed. The output of the amplifier data will be directed to a computer with BrainVision Pycoder software to record the obtained records and the data will be processed using the BrainVision Analyzer.
Motor aspects of daily life | Baseline, after 6 weeks, and after 10 weeks
  The Unified Parkinson's Disease Assessment Scale - Part II (MDS-UPDRS) will be used to assess the motor experiences of daily life.
Stroop test | Baseline, after 6 weeks, and after 10 weeks
  A modified version of the Stroop Test will be used, the Victoria Stroop Test (VST), which uses three conditions: name the color 24 points, 24 neutral words and 24 colorful words printed in incongruous colors.
Dual Task | Baseline, after 6 weeks, and after 10 weeks
  Participants will perform single and double task conditions with Timed Up and Go (TUG). First, only TUG (TUGS) is performed, a single attention task in which the participant will be instructed to get up from a chair, walk at a normal and safe pace for three meters, rotate 180 degrees, come back and sit down. Then the TUG will be performed simultaneously performing the cognitive task of generating a word list starting with a specific letter, speaking out loud (TUGC), and performing the TUG with the motor task of carrying a glass of water ( TUGM).
Verbal Fluency Test | Baseline, after 6 weeks, and after 10 weeks
  The FAS is a verbal fluency test, in which participants must name as many unique words as possible starting with the letters F, A and S in separate tests, and each condition has a time limit of 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraiba
Locations (1):
- Suellen Marinho Andrade, João Pessoa, Paraíba, Brazil